CLINICAL TRIAL: NCT06662357
Title: Family Connections: A Community-Based Approach to Expanding Mental Health Access and Engagement for SED Youth
Brief Title: Family Connections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Responsible Party: Principal Investigator, Katherine Grimes MD, Children's Health Initiative, Director, Cambridge Health Alliance
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H79SM089682; H79SM089682 (Other Grant/Funding Number: SAMHSA)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Emotional Disturbance; Behavior Disorders in Children
MeSH Terms: conditions — Affective Symptoms; Child Behavior Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: The Family Connections Model consists of the delivery of intensively integrated clinical care within pediatrics, combined with community-based parent support from family support specialists. Innovations include child mental health specialists joining the pediatrics team for "huddles", psychiatry notes shared with pediatricians via the Electronic Medical Records and active inclusion of pediatricians in pre-evaluation discussions with the Family Connections Team and post-evaluation recommendations for the families. In addition, the Safety-Net model includes active communication with school personnel, child welfare, and community-based resources, when needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator: Family Connections Intervention (Active Comparator)
  Interventions: Behavioral: Behavioral Treatment
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Behavioral Treatment — "Family Connections" Care Planning Team: Clinical expertise will be combined with peer-to-peer parent/guardian support for trauma-informed care delivery to both parent and child. All aspects of the care continuum will be provided in a culturally and linguistically competent manner, with child and family-driven care planning.
  Arms: Active Comparator: Family Connections Intervention

SUMMARY:
The Family Connections study, is intended to disrupt disparities in mental health treatment access for children at-risk for childhood trauma (ACEs) and/or serious emotional disturbance (SED). "Family Connections" will use mobile clinical and family support teams to improve mental health outcomes. This clinical innovation, nested in an integrated system-of-care will be piloted for children, ages 3-18 yrs., with SED who receive primary care through Cambridge Health Alliance.

ELIGIBILITY:
Inclusion Criteria:

* 3 through 18 years (17½ years maximum at time of enrollment)
* Referred by Primary Care Physician's (PCP) from one of the three Cambridge Health Alliance (CHA) primary care intervention sites to the Family Connections team for an integrated child mental health and/or substance use disorder clinical assessment.
* Positive screen on CHA's standard pediatric mental health and substance use screening instruments, and/or parental concern about possible mental health/substance use needs, and/or PCP concern about possible mental health/substance use needs
* Enrolled in MassHealth

Exclusion Criteria:

* Subjects over 17.5 years (SAMHSA data collection required at 6 and 12 months after enrollment which must occur before age 18 years.)
* Youth who are not enrolled in MassHealth
* CHA patients with PCP located at CHA primary care site other than the identified intervention sites

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Changes in Child and Adolescent Functional Assessment Scale (CAFAS) Score | Baseline collected at enrollment, follow-up assessments collected at 6 months and 12 months
  Comparative analysis of baseline and follow-up clinical functioning scores
  CAFAS Scoring:
  Levels of Dysfunction None or minimal 0-10 Mild 20-30 Moderate 40-60 Marked 70-80 Severe >90
Changes in Children's Global Assessment Scale (CGAS) Score | Baseline collected at enrollment, follow-up assessments collected at 6 months and 12 months
  Comparative analysis of baseline and follow-up clinical functioning scores
  CGAS Scale:
  100-91 Superior functioning 90-81 Good functioning 80-71 No more than a slight impairment in functioning 70-61 Some difficulty in a single area, but generally functioning pretty well 60-51 Variable functioning with sporadic difficulties 50-41 Moderate degree of interference in functioning 40-31 Major impairment to functioning in several areas 30-21 Unable to function in almost all areas 20-11 Needs considerable supervision 10-1 Needs constant supervision
Family perceptions of care using the Family Professional Partnership Scale (FPPS). | Baseline collected at enrollment, follow-up assessments collected at 6 months and 12 months
  Analysis of baseline and follow-up family perceptions of care (18 Questions):
  1. - Very Dissatisfied
  2. - Dissatisfied
  3. - Neither
  4. - Satisfied
  5. - Very Satisfied
Access to child mental health and substance abuse (MH/SA) care | 0-6 months
  Comparative analysis of access to care trends
Engagement in child mental health and substance abuse (MH/SA) treatment | 6-12 months
  Comparative analysis of service use trends

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Grimes, MD, MPH, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States